CLINICAL TRIAL: NCT02924116
Title: Use of Bioboosti Non-pharmacologic Device for Insomnia Treatment: A Pilot Study
Brief Title: Bioboosti Device for Insomnia Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Biomobie (Unknown); Harvard University (Other)
Responsible Party: Principal Investigator, Pavlova, Milena,M.D., Medical Doctor, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000996
Record Dates: First submitted 2016-09-20; First posted 2016-10-05 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Insomnia
Keywords: insomnia; sleep; Bioboosti; Biomobie; device
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Subjects will complete the first arm of the study. Upon completion, the subjects will be offered enrollment into the next long term arm of the study (Sustained Efficacy).
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bioboosti (Experimental): Treatment with the Bioboosti device for two weeks. The device produces a pulsed micro-magnetic field. Subjects will use it once a day for about one hour, before habitual sleep time.
  Interventions: Device: Bioboosti
- Sustained Efficacy (Experimental): Treatment with Bioboosti device for a year. In order to see if the device has sustained efficacy in treating insomnia.
  Subjects will use it once a day for about one hour, before habitual sleep time.
  Interventions: Device: Bioboosti
- Insomnia and migraine (Experimental): Treatment with the Bioboosti device for a month. Subjects will use it once a day for about one hour, before habitual sleep time.
  Interventions: Device: Bioboosti

INTERVENTIONS:
Device: Bioboosti — Subjects will place the device on the palm of their hand for 8 minutes. There is a light on the device that changes to indicate that the 8 minutes have passed. They will then place it on the palm of the other hand and keep it there for 8 minutes. Alternating 8-minute cycles between hands will be done up to 6 times.

SUMMARY:
The purpose of this study is to determine the effects of the Bioboosti device on sleep for patients who have been diagnosed with insomnia.

DETAILED DESCRIPTION:
Insomnia is a common health complaint that is associated with discomfort, loss of productivity, poor health and higher use of healthcare. The use of non-pharmacologic treatments for insomnia has gained much attention in recent years. The investigators are conducting this research because a safe, non-pharmacologic treatment would benefit patients with insomnia, and to see if the Bioboosti device is an effective treatment for insomnia.

Subjects will include patients from the clinics who have the diagnosis of insomnia. Study staff will notify the treating physician of a potential subject. If the subject gives permission and would like to obtain more information, study staff will approach them and provide them with the consent form to review. Study staff may also contact them by phone to explain the study and recruit.

Subjects will be asked to make 5 visits:

Visit 1-- consent form, physical exam, vitals, pregnancy test, sleep log

Visit 2-- sleep questionnaires, urine test for hormones associated with sleep, sleep log, placement of EEG

Visit 3-- remove EEG, beginning of treatment with Bioboosti device, sleep log Treatment phase-- subjects use the Bioboosti at home for two weeks

Visit 4-- return of Bioboosti, sleep questionnaires, urine test for hormones associated with sleep, sleep log, placement of EEG

Visit 5-- remove EEG, collect sleep logs

ELIGIBILITY:
Inclusion Criteria:

* Patients with insomnia

Exclusion Criteria:

* Untreated moderate or severe sleep apnea
* Major circadian rhythm disorder
* Pregnant women
* Breastfeeding
* Cardiac pacemaker
* Cancer
* Severe conditions related to heart, brain, kidney and hematopoietic system
* Severe/unstable angina pectoris
* Arteria coronaria/ peripheral arterial bypass graft
* Acute congestive heart failure
* Renal insufficiency
* Mechanical intestinal obstruction
* Any electrical devices

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2024-11 (Actual); Study Completion 2025-04 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia symptoms before treatment to after treatment | Week 1, Week 4
  Within subject comparisons before and after treatment, subjects answer questions on their sleep habits.
Change in Sleepiness before treatment to after treatment | Week 1, Week 4
  Within subject comparisons before and after treatment, subjects answer questions on sleep difficulty.

SECONDARY OUTCOMES:
Change in EEG from before treatment to after treatment | Week 2, Week 4
  Ambulatory EEG will be used before treatment and after treatment, using sleep montage per standard AASM criteria and scored by a registered polysomnography technologist using AASM guidelines. Sleep architecture will be reported as the percent of time the subject remains in the different sleep stages. Specifically we will compare percent in REM sleep before and after treatment. The waveform of the EEG that will be assessed during teh study period is delta.

CONTACTS AND LOCATIONS:
Overall Officials: Milena Pavlova, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT02924116/Prot_SAP_001.pdf
  • Informed Consent Form (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT02924116/ICF_000.pdf